CLINICAL TRIAL: NCT04166500
Title: Early Outpatient Hysteroscopy Can Prevent Intrauterine Adhesion After Induced Abortion: a Randomized Controlled Trial
Brief Title: Early Outpatient Hysteroscopy Can Prevent Intrauterine Adhesion After Induced Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CMRPG8J1131
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hysteroscopy; Intrauterine Adhesion
Keywords: Induced abortion; Uterine adhesions; Reproductive infertility; Hysteroscopy
MeSH Terms: conditions — Gynatresia | interventions — Hysteroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Procedure: Hysteroscopy
- Control (No Intervention)

INTERVENTIONS:
Procedure: Hysteroscopy — outpatient hysteroscopy after the first menstrual cycle in the follicular phase (9-12 days).
  Arms: Intervention

SUMMARY:
Background: Intrauterine adhesions are a difficult clinical problem for reproductive infertility. The most common cause is uterine cavity surgery and post-abortion (including abortion and spontaneous abortion). After the abortion, the uterine cavity adhesion, when is the key point, the literature is not much ink, early literature has mentioned that after the abortion, the uterus scraping action is scraped in four days and the uterine adhesion will be smaller than one to four weeks. Much more, it seems that the sooner the uterine adhesion factor is excluded, the more it can reduce uterine adhesion, but the uterine curettage itself is a risk factor for uterine adhesion. This early practice, the current clinical application, is not used, Instead, it is a hysteroscopy. Our past clinical observations, as soon as possible after the abortion, outpatient hysteroscopy, can find the tissue factors that may cause adhesion in the uterine cavity as soon as possible, and immediately remove it with an outpatient hysteroscope.

Objective: To verify the early outpatient hysteroscopy and reduce the occurrence of intrauterine adhesion after abortion.

Expected benefits to patients: Abortion is likely to cause intrauterine adhesions, which may further cause the incidence of reproductive infertility, should be involved before the formation of permanent injury, reduce the adhesion of the uterine cavity. Outpatient hysteroscopy is a simple and easy-to-use examination procedure that is painless and does not require anesthesia. Although it is invasive but has few complications, it is expected to reduce the occurrence of intrauterine adhesion after abortion.

ELIGIBILITY:
Inclusion Criteria:

* female age 20 to 45 years-old
* undergo induced abortion
* desire future fertility
* agree with the trial and sign the consent form

Exclusion Criteria:

* previous intrauterine surgery
* previous intrauterine adhesion
* previous having over(and/or equal to) 3 times of induced abortion
* infection condition

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence rate of intrauterine adhesions | 6 months later after induced abortion
  assess with hysteroscopy

SECONDARY OUTCOMES:
The American Fertility Society (AFS) intrauterine adhesion (IUA) score | 6 months later after induced abortion
  Assess by hysteroscopy and measure with IUA score. Score scaling from 1 to 12 with the higher scores mean a worse outcome. Stage I (mild, 1-4), stage II (moderate, 5-8); stage III (severe, 9-12).
Menstrual cycle condition: Menstrual amount | 6 months later after induced abortion
  Normal/Hypo/Hyper by Pictorial blood loss assessment charts (PBACs): self-reported by patients and questionnaire.
  Normal amount: 10 to 100 points. Hypermenorrhea: over 100 points. Hypomenorrhea: less than 10 points.
Menstrual cycle condition: Menstrual duration | 6 months later after induced abortion
  days: by questionnaire
Menstrual cycle condition: Menstrual symptoms | 6 months later after induced abortion
  dysmenorrhea/no dysmenorrhea: by questionnaire
Sonography findings:endometrial thickness | 6 months later after induced abortion
  centimeters
Sonography findings: morphology | 6 months later after induced abortion
  Normal. Abnormal (hyperechogenic lesion/hypoechogenic lesion/other irregular endometrial line)
Fertility outcome | 2 years later after induced abortion
  Pregnancy outcome: no pregnancy/ abortion/ gestational age/ live birth

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsai NC, Hsiao YY, Su YT, Lin YJ, Kung FT, Chen PH, Lan KC. The efficacy of early office hysteroscopy in preventing intrauterine adhesions after abortion: a randomized controlled trial. BMC Womens Health. 2024 Jul 13;24(1):400. doi: 10.1186/s12905-024-03247-0. PMID 39003483